CLINICAL TRIAL: NCT02552381
Title: Evaluation of Fibrin Structure Marker in Cancer Patients Treated and Not Treated With LMWH
Acronym: FICT
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago R&D (Industry)
Collaborators: Hôpital Louis Mourier (Other); Hopital Lariboisière (Other)
Responsible Party: Sponsor
Other Study IDs: FICT 2015-A00501-48
Record Dates: First submitted 2015-08-13; First posted 2015-09-17 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Malignant Tumor
Keywords: Cancer; Thromboembolic event; Fibrin Structure; LMWH
MeSH Terms: conditions — Neoplasms; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen citrated Poor Platelets Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group I: Patients without LMWH treatment.
  A thromboembolic event has to be diagnosed according to standard imaging criteria (spiral computed tomography CT, proximal lower limb venous compression ultrasonography US) by clinicians who will not have knowledge of the result of the fibrin structure marker.
  The following assays will be performed for these patients :
  * Fibrin Structure measured at baseline and every month using prototype assays
  * Other markers activity : sFVIII:C and TFPI for coagulation activation, DDimers and PAI-1 for fibrinolysis resistance and fibrin assay, all measured at baseline and every 3 months.
  Interventions: Other: Fibrin Structure
- Group II: Patients with LMWH treatment at prophylactic dose at enrollment only.
  A thromboembolic event has to be diagnosed according to standard imaging criteria (spiral computed tomography CT, proximal lower limb venous compression ultrasonography US) by clinicians who will not have knowledge of the result of the fibrin structure marker.
  The following assays will be performed for these patients :
  * Fibrin Structure measured at baseline and every month using prototype assays,
  * Anti-FXa activity measured at baseline and every month,
  * Other markers activity : FVIII:C and TFPI for coagulation activation, DDimers and PAI-1 for fibrinolysis resistance and fibrin assay, all measured at baseline and every 3 months.
  Interventions: Other: Fibrin Structure
- Group III: Patients with LMWH treatment at therapeutic dose.
  A thromboembolic event has to be diagnosed according to standard imaging criteria (spiral computed tomography CT, proximal lower limb venous compression ultrasonography US) by clinicians who will not have knowledge of the result of the fibrin structure marker.
  The following assays will be performed for these patients :
  * Fibrin Structure measured at baseline and every month using prototype assays,
  * Anti-FXa activity measured at baseline and every month,
  * Other markers activity : FVIII:C and TFPI for coagulation activation, DDimers and PAI-1 for fibrinolysis resistance and fibrin assay, all measured at baseline and every 3 months.
  Interventions: Other: Fibrin Structure

INTERVENTIONS:
Other: Fibrin Structure — Modifications of Fibrin Structure in patients who have developed VTE in comparison with patients without VTE.

SUMMARY:
The purpose of the study is to assess the fibrin structure marker in the plasma of cancer patients, treated or not treated with LMWH at prophylactic or therapeutic doses, in order to determine the venous thromboembolic risk. The occurrence of thromboembolic events in patients without treatment and in patients under LMWH treatment will be recorded, depending on the location and type of cancer, metastases, and treatment of cancer.

DETAILED DESCRIPTION:
Rationale. Venous thromboembolism (VTE) is a major complication often encountered in oncology and onco-hematology, and difficult to handle. It involves the activation of coagulation with the generation of fibrin and plasmin and angiogenesis activation. Low molecular weight heparins (LMWH) are used to treat cancer associated thrombosis. Furthermore, they could have an inhibitory effect on tumor progression.

International recommendations on the treatment and prophylaxis of the disease allow a better management of VTE in patients with cancer. Its prevalence is high, occurring in 15-20% of the patients. It remains the second leading cause of death after cancer. LMWH at therapeutic dosage for at least three months and preferably six months without oral bridging is the reference treatment for VTE, which showed a 50% reduction in the risk of recurrent thromboembolism without increasing the hemorrhagic risk. In case of VTE recurrence under LMWH treatment, the dose can be increased by 10%. Preliminary results suggest that the fibrin structure marker would predict the hemorrhagic or thromboembolic risk, and show that LMWH has a dose-dependent effect on fibrin structure. This marker is evaluated as a tool to guide the treatment of VTE by LMWH in patients with cancer.

Main objective. To assess the fibrin structure marker in the plasma of cancer patients, treated or not treated with LMWH at prophylactic doses at enrollment or therapeutic doses, to determine the venous thromboembolic risk. The occurrence of thromboembolic events in patients without treatment or of recurrent thromboembolic events in patients under LMWH treatment will be studied, depending on the location and type of cancer, metastases, and treatment of cancer.

Patients. At least 300 adult patients over 18 years with all types of malignancies documented before or during therapeutic treatment with LMWH for thromboembolic event. They will be monitored every month in consultation or during hospitalization in the Internal Medicine Department. The patients under prophylaxis with LMWH at enrollment will also be included and classified in the group of prophylactic patients. The patients who receive prophylactic treatment during will be included and classified in the group of untreated patients.

Will not be included: patients with sepsis, severe infections, pneumonia, surgery, suspected thromboembolic event related to catheter implantation, vitamin K antagonists (VKA) in progress, and those with impossible follow-up.

The study is conducted in compliance with French regulation after ethics approval, the authorization for processing personal data (Commission Nationale de l'Informatique et des Libertés, 8, rue Vivienne CS 30223 75083 Paris Cedex 02) receipt number 1867686 v 0, date 18 June 2015.

Reference algorithm. Patients will be supported for the diagnosis and specific treatment of cancer (with or without metastases), according to the daily practice. The baseline risk score is the Khorana score of clinical probability, based on clinical criteria. A thromboembolic event has to be diagnosed according to standard imaging criteria (spiral computed tomography CT, proximal lower limb venous compression ultrasonography US) by clinicians who will not have knowledge of the result of the fibrin structure marker.

Biological parameters to be studied. The following tests will be carried out on frozen citrated plasma or serum, without knowledge of the clinical data and the conclusion of a diagnostic of thromboembolic event:

* Structure of the fibrin using coag-lysis method, measured at baseline and every month for all patients, by one site, using prototype assays
* Anti-FXa activity measured at baseline and every month only for patients treated with LMWH at therapeutic doses,
* FVIII:C and TFPI for coagulation activation, DDimers and PAI-1 for fibrinolysis resistance, Fibrin assay for inflammation and hypercoagulation evaluation, all measured at baseline and every 3 months for all patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-opposition to participate in the evaluation
* patients from Internal Medicine Department
* patients affected with all types of malignancies, treated or not with LMWH

Exclusion Criteria:

* patients treated with VKA or with recent surgery (within one month)
* patients with a condition known to cause a coagulation activation status other than cancer (sepsis, pneumonia,..)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Internal Medicine Department, in a French Hospital
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2015-08; Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Dynamic evolution of the optical density delta (ODD) | 36 Months
  Evolution of the optical density delta (ODD) and temporal parameters in patients who have developed VTE in comparison with those without VTE; variations of the Fibrin Structure parameters in comparison with either coagulation activation or fibrinolysis resistance assays, or fibrin assay.
  Changes of the Fibrin structure parameters in patients of group III in comparison with group I and/or group II.

SECONDARY OUTCOMES:
Clotting time (s) | 36 Months
  Evolution of the optical density delta (ODD) and temporal parameters in patients who have developed VTE in comparison with those without VTE; variations of the Fibrin Structure parameters in comparison with either coagulation activation or fibrinolysis resistance assays, or fibrin assay.
  Changes of the Fibrin structure parameters in patients of group III in comparison with group I and/or group II.
Fibrin formation time (s) | 36 Months
  Evolution of the optical density delta (ODD) and temporal parameters in patients who have developed VTE in comparison with those without VTE; variations of the Fibrin Structure parameters in comparison with either coagulation activation or fibrinolysis resistance assays, or fibrin assay.
  Changes of the Fibrin structure parameters in patients of group III in comparison with group I and/or group II.
Lysis time (s) | 36 Months
  Evolution of the optical density delta (ODD) and temporal parameters in patients who have developed VTE in comparison with those without VTE; variations of the Fibrin Structure parameters in comparison with either coagulation activation or fibrinolysis resistance assays, or fibrin assay.
  Changes of the Fibrin structure parameters in patients of group III in comparison with group I and/or group II.
Duration and level of the plateau (s) | 36 Months
  Evolution of the optical density delta (ODD) and temporal parameters in patients who have developed VTE in comparison with those without VTE; variations of the Fibrin Structure parameters in comparison with either coagulation activation or fibrinolysis resistance assays, or fibrin assay.
  Changes of the Fibrin structure parameters in patients of group III in comparison with group I and/or group II.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mahe, MD, PhD, Principal Investigator — Université of Paris 7 - Paris Diderot; Geneviève Contant, PhD, Study Director — Diagnostica Stago
Locations (1):
- Internal Medecine Department - Adults Pole and Hematology Laboratory Hôpital Louis Mourier (AP-HP), Colombes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meyer G. [Looking for the best molecule. A short history of anticoagulants]. Rev Mal Respir. 2011 Oct;28(8):951-3. doi: 10.1016/j.rmr.2011.09.006. Epub 2011 Oct 15. No abstract available. French. PMID 22099399
- [Background] Campbell RA, Aleman M, Gray LD, Falvo MR, Wolberg AS. Flow profoundly influences fibrin network structure: implications for fibrin formation and clot stability in haemostasis. Thromb Haemost. 2010 Dec;104(6):1281-4. doi: 10.1160/TH10-07-0442. Epub 2010 Sep 30. No abstract available. PMID 20886193
- [Background] Wolberg AS, Gabriel DA, Hoffman M. Analyzing fibrin clot structure using a microplate reader. Blood Coagul Fibrinolysis. 2002 Sep;13(6):533-9. doi: 10.1097/00001721-200209000-00008. PMID 12192305
- [Background] Varin R, Mirshahi S, Mirshahi P, Kierzek G, Sebaoun D, Mishal Z, Vannier JP, Yvonne Borg J, Simoneau G, Soria C, Soria J. Clot structure modification by fondaparinux and consequence on fibrinolysis: a new mechanism of antithrombotic activity. Thromb Haemost. 2007 Jan;97(1):27-31. PMID 17200767
- [Background] Pieters M, Philippou H, Undas A, de Lange Z, Rijken DC, Mutch NJ; Subcommittee on Factor XIII and Fibrinogen, and the Subcommittee on Fibrinolysis. An international study on the feasibility of a standardized combined plasma clot turbidity and lysis assay: communication from the SSC of the ISTH. J Thromb Haemost. 2018 May;16(5):1007-1012. doi: 10.1111/jth.14002. Epub 2018 Apr 15. No abstract available. PMID 29658191
- [Background] Longstaff C; subcommittee on fibrinolysis. Development of Shiny app tools to simplify and standardize the analysis of hemostasis assay data: communication from the SSC of the ISTH. J Thromb Haemost. 2017 May;15(5):1044-1046. doi: 10.1111/jth.13656. Epub 2017 Mar 17. No abstract available. PMID 28304129
- See also: Recommandations internationales pour le traitement et la prophylaxie de la thromboembolie veineuse chez le patient cancéreux. GFTC, Communiqué de presse, 26 Juin 2013 — http://www.thrombose-cancer.com/
- See also: Patent : Juillet 2015, Method for determining the structural profile of a fibrin clot reflecting the stability thereof, in order to predict the risk of bleeding, thrombosis or rethrombosis — https://patentscope.wipo.int/search/fr/detail.jsf?docId=WO2016012729&redirectedID=true